CLINICAL TRIAL: NCT01515878
Title: Hemocontrol's Effectiveness in a RAndomized Controlled Trial on the Reduction of Cardiovascular Long-term EventS
Brief Title: Hemocontrol's Effectiveness on the Reduction of Cardiovascular Long-term EventS
Acronym: HERACLES
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Antonio Santoro, Professor, MD, Chief of Nephrology, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Kidney Failure Chronic; Cardiovascular Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dialysis with BVT (Experimental): Dialysis using the BVT monitor biofeedback called Hemocontrol
  Interventions: Device: Hemocontrol
- Conventional dialysis (No Intervention): Conventional dialysis without blood volume tracking or similar therapies

INTERVENTIONS:
Device: Hemocontrol — Blood Volume Tracking system using biofeedback
  Arms: Dialysis with BVT

SUMMARY:
It is hypothesized that a consistent use of the Hemocontrol TM biofeedback function improves long-term cardiovascular outcome, mediated by reduced hypertension due to fluid overload and by reduced incidence of intradialytic hypotensive episodes

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 65 years old
2. Arterial Hypertension: predialysis SBP >140 mmHg and/or DBP >90 mmHg in at least 50% over the previous month dialysis sessions or receiving at least one antihypertensive pharmacological drug including diuretics, disregarded blood pressure value
3. On a three times per week hemodialysis schedule
4. Time on hemodialysis less than 6 months
5. Able to measure their blood pressure at home (by themselves or with the aid of the care giver)
6. Signed informed consent

Exclusion Criteria:

1. Active neoplastic disease
2. Mental illness
3. Pregnancy
4. Single needle treatment
5. Inability, as judged by the investigator, to follow or understand the protocol instructions
6. Blood flow rate less than 200 mL/min
7. Patients who at the time of recruitment need clinical indication for special renal replacement therapies and/or on treatment with one of the following modalities: HDF or similar diffusive-convective therapies, treatment time >5h, blood temperature control, isolated UF profiling of Na/UFR
8. Patients with a life expectancy shorter than 6 months
9. Patients in a list for transplant within the next 6 months
10. Predialysis Hemoglobin level greater than 13.5 g/dl
11. History of major cardiovascular events during run in period

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 36 months
  The primary objective will be assessed by the incidence rate of Fatal and not fatal cardiovascular events

SECONDARY OUTCOMES:
Cardiovascular morbidity | 36 months
  * Number of hospital admissions evaluated as annual hospitalization rate related to: Non fatal myocardial infarction, New-onset angina, Non fatal stroke, Congestive heart failure, Transient ischemic attack, Pulmonary oedema
  * Length of stay during hospitalization;
  * Number of extra dialysis or prolonged dialysis due to fluid overload.
Blood pressure control | 36 months
  Blood pressure control:
  * Predialysis blood pressure measurements
  * Home blood pressure self assessment
  * Antihypertensive therapy changes
  * Proportion of patients achieving adequate blood pressure control
  * Intradialytic acute hypotension:
Quality of life and dialysis tolerance evaluated with questionnaire. | 36 months
  Questions of the KDQOL36 questionnaire
Dry weight management | 36 months
  Optional when available at site: Hydration status estimated by Cardiothoracic index or BNP or BIA at baseline and each 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mac Rae, MD, Study Chair — Calgary hospital, Canada; Hafedh Fessi, MD, Study Chair — APHP Tenon, Paris France; Juan Buades, MD, Study Chair — Majorca hospital, Spain; Helena Mancini, MD, Study Chair — AOSP, Bologna Italy; Antonio Santoro, Pf, Study Chair — AOSP, Bologna Italy
Locations (3):
- Health Regional hospital, Calgary, Canada
- Hopital Tenon, APHP, Paris, France
- Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy